CLINICAL TRIAL: NCT05474677
Title: The Suture Size in Laparotomy Wound Closure to Prevent Post-operative Complications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Raya Al shaaibi (Other Government)
Responsible Party: Sponsor-Investigator, Raya Al shaaibi, Dr, Oman Medical Speciality Board
Organization: Oman Medical Speciality Board (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OmanMedSB
Record Dates: First submitted 2022-07-23; First posted 2022-07-26 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Suture Size, Incisional Hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): intervention group with the abdomen will be closed with continuous PDS 2\0 sutures
  Interventions: Procedure: closure of the abdominal fascia
- control group (Experimental): the abdomen will be closed with continuous sutures size zero
  Interventions: Procedure: closure of the abdominal fascia

INTERVENTIONS:
Procedure: closure of the abdominal fascia — The abdomen will be closed in intervention group with continuous PDS 2\0 sutures and size zero in control group.

SUMMARY:
Background: Incisional hernia is a common complication of midline laparotomy, and it is associated with high morbidity and high costs. Suture size used in the closure of the abdominal wall fascia was not studied independently.

Objective: Identify the best suture size for closure of the fascia following laparotomy incisions, by assessing the suture size 2\0 versus zero.

Research methods: Prospective, multicentric, randomized controlled and double-blind trial. Patients undergoing elective or emergency laparotomy in Royal Hospital, Sultan Qaboos University Hospital and Armed Force Hospital between 2022 and 2023. We aimed for a total of 276 patients (n=138 per group). The abdomen will be closed in intervention group with continuous PDS 2\0 sutures and size zero in control group. Patients will be followed for immediate post-operative wound complications and late complication after 6 months then after one year.

DETAILED DESCRIPTION:
Objectives and hypothesis of the study The primary objective: to identify the best suture size for closure of the fascia following laparotomy incisions to prevent incisional hernia, by assessing the suture size 2\0 versus zero.

Secondary objective: assess the incidence of wound dehiscence and wound infection in two studied group.

Study hypothesis: Suture size 2/0 decreases the incidence of incisional hernia in the closure of the abdominal fascia

Research design and Methods Study design: Prospective, multicentric, randomized controlled and double-blind trial.

Characteristics of study area and target population Patients undergoing elective or emergency laparotomy in Royal Hospital, Sultan Qaboos University Hospital and Armed Force Hospital between 2022 and 2023. Eligible patients are adults aged 18 years or older, who signed informed consent and the expected survival more than one year. Patients with history of midline laparotomy within 3 months, pregnant patients and patients with history of incisional hernia will be excluded from the study.

Sampling we estimated that 125 patients would be needed in each group to provide 80% power to detect a reduction of at least 50% (18% in the classic group vs 6% in the 2.0 group) in the incidence of incisional hernia at a two-sided alpha level 0.05. We aimed for a total of 276 patients (n=138 per group) to correct for an estimated 10% loss to follow-up in each group. The statistical method used was Fisher's exact test. The calculation was done using the software G*Power version 3.1.9.2. Randomization will be achieved by using a software.

Variable definitions and measurements The abdomen will be closed in the intervention group patients with continuous PDS 2\0 sutures, half centimeter between each stitch. The control group will be closed by the conventional method in the Royal Hospital, continuous using double-looped. Sex, age, BMI, smoking, diabetes mellitus, COPD, cardiovascular disease, corticosteroid use, previous laparotomy, ASA classification, preoperative chemotherapy, preoperative radiotherapy, type of surgery are the variable which will be studied.

Data collection tools and methods Data will be entered using Epi-data software.

Data quality State how data will be entered using Epi-data software.

Data analysis Continuous variables will be presented as mean, median, and standard deviation whereas, categorical variables will be presented as frequency and percentage. Comparison of means between two groups will be assessed using the independent samples t-test or the Mann-Whitney U test, as appropriate. Association between two categorical variables will be assessed using an appropriate Chi-square test (Likelihood ratio test or Fisher's exact test). Multivariate log-binomial regression analysis will be used to determine the independent risk factors for the development of incisional hernia. A P-value less than 0.05 will be considered statistically significant. All the analysis will be done using the IBM SPSS statistics version 26.0.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 years or older, who signed informed consent and the expected survival more than one year.

Exclusion Criteria:

* Patients with history of midline laparotomy within 3 months, pregnant patients and patients with history of incisional hernia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
incisional hernia | 6 months and one year
  development of incisional hernia post operative

SECONDARY OUTCOMES:
wound infection | 30 days
  development of wound infection post operative
wound dehiscence | 30 days
  development of wound dehiscence post operative

CONTACTS AND LOCATIONS:
Overall Officials: mohmmed al abri, consultant, Study Director — Oman Medical Specialty Board
Locations (1):
- Raya Al Shaaibi, Muscat, Oman

IPD SHARING:
Plan to Share IPD: No
participant data will not be shared